CLINICAL TRIAL: NCT02332239
Title: Text-Message-Based Depression Prevention for High-Risk Youth in the ED
Acronym: iDOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23MH095866 (NIH); K23MH095866 (NIH)
Record Dates: First submitted 2014-12-29; First posted 2015-01-06 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Depressive Disorder; Violence
Keywords: depression; violence; emergency department; mhealth; text message
MeSH Terms: conditions — Depressive Disorder; Depression; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iDOVE Intervention (ED+text) (Experimental): 1. In-ED brief session, introducing basic principles of cognitive behavioral theory and the structure of the text-message portion of the intervention
  2. Eight-week longitudinal tailored CBT-based text-message program
  Interventions: Behavioral: iDOVE Intervention (ED+text)
- Control (EUC) (Placebo Comparator): 1. In-ED brief session, discussing home safety & nutrition
  2. Eight-week longitudinal home safety & nutrition text-message program
  Interventions: Behavioral: Control (EUC)

INTERVENTIONS:
Behavioral: iDOVE Intervention (ED+text) — 1. In-ED brief session, introducing basic principles of cognitive behavioral theory and the structure of the text-message portion of the intervention
  2. Eight-week longitudinal tailored text-message program
  Arms: iDOVE Intervention (ED+text)
Behavioral: Control (EUC) — 1. In-ED brief session, discussing home safety & nutrition
  2. Eight-week longitudinal home safety & nutrition text-message program
  Arms: Control (EUC)

SUMMARY:
The purpose of this randomized controlled study is to evaluate acceptability and feasibility, and to gather preliminary data about efficacy, of "iDOVE," a brief emergency department introductory session + longitudinal automated text-message depression prevention program for high-risk teens.

DETAILED DESCRIPTION:
Peer violence and depressive symptoms have mutual, reinforcing negative impacts on teens' emotional and behavioral regulation strategies.

The emergency department (ED) is the primary source of care for many high-risk teens. It provides an opportunity to initiate preventive interventions, to complement existing mental health treatment or to stand alone for those who may lack access to formal care. Personalized text-message interventions are accessible, feasible, and may be effective with these adolescents.

The purpose of this study is to test the feasibility and acceptability of a novel text-message augmented depression prevention intervention, "iDOVE." Drawing on effective cognitive behavioral therapy (CBT) and motivational interviewing (MI) depression and violence prevention interventions, a brief in-ED session will introduce basic cognitive and behavioral strategies. Following ED discharge, eight weeks of tailored CBT-informed daily text messages will be sent, to enhance skills and remind participants of self-determined goals.

Participants will be identified in the course of usual ED care. If eligible, parents will be consented and participants assented. Participants will complete a baseline assessment and will be randomized to experimental (ED+text, n=50) or enhanced usual care (EUC, n=50) care, using stratified block randomization.

ED+text group participants will participate in a brief, structured in-ED introduction on CBT and the iDOVE program, followed by 8 weeks of tailored, two-way, CBT-and MI-informed automated text messages (short message service, SMS). EUC group participants will participate in a brief, structured, in-ED introduction to home safety & nutrition, followed by 8 weeks of automated SMS regarding home safety & nutrition. The current standard of care for these patients is no care: no depression or violence screening assessment protocols are currently used in our ED. Both ED+text and EUC conditions therefore exceed current levels of care.

At baseline, 8 week follow-up, and 16 week follow-up, participants will complete assessments on depressive symptoms, violence, cognitive/behavioral skill-sets, and resource utilization. At the 8-week follow-up, standardized qualitative and quantitative process measures will be administered to assess efficacy, acceptability, usability, and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* presenting to the emergency department for routine care
* reporting past-year physical violence (using a modified version of The Revised Conflict Tactics Scales (CTS)) and current mild-to-moderate depressive symptoms (using Patient Health Questionnaire (PHQ)-9), as identified on a brief screen administered in the ED
* accompanied by a consentable parent
* own or have access to a text-message-capable mobile phone

Exclusion Criteria:

* medically/physically unable to assent
* chief complaint of suicidal ideation, psychosis, or child abuse
* in police custody
* severe depressive symptoms

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ranney, MD MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital Emergency Department, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Less than 150 randomized controlled trial (RCT) participants

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1,190 potential screening subjects presenting to the ED for any reason during from February-December 2015, 1063 consented to screening. Of these, 1031 were successfully screened and 142 met eligibility criteria for the full trial. Of those eligible for the full randomized controlled trial (RCT), 116 consented.
Groups:
- iDOVE Intervention (ED+Text): 1. In-ED brief session, introducing basic principles of cognitive behavioral theory and the structure of the text-message portion of the intervention
  2. Eight-week longitudinal tailored CBT-based text-message program
  iDOVE Intervention (ED+text): 1) In-ED brief session, introducing basic principles of cognitive behavioral theory and the structure of the text-message portion of the intervention 2) Eight-week longitudinal tailored text-message program
- Control (EUC): 1. In-ED brief session, discussing home safety & nutrition
  2. Eight-week longitudinal home safety & nutrition text-message program
  Control (EUC): 1) In-ED brief session, discussing home safety & nutrition 2) Eight-week longitudinal home safety & nutrition text-message program
Period: Overall Study
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
Started | 58 | 58
Completed | 54 | 52
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC) | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.83 (1.23) | 15.05 (1.13) | 14.94 (1.18)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 34 | 34 | 68
  Gender: Male | 24 | 22 | 46
  Gender: Transgender, Other, Prefer not to answer | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 23 | 41
  Not Hispanic or Latino | 39 | 35 | 74
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 5 | 2 | 7
  White | 29 | 28 | 57
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 116
School Year [Count of Participants; unit: Participants]
  Grades 6-8 | 16 | 10 | 26
  Grades 9-12 | 37 | 48 | 85
  College | 2 | 0 | 2
  Not in school | 3 | 0 | 3
Socio-economic status [Count of Participants; unit: Participants] — Socioeconomic Status (SES) was collected using selected items from the National Study for Adolescent Health. "Low" SES was defined as receipt of free services (a parent or guardian who qualifies for public assistance, welfare, food stamps, disability benefits, Medicaid, Rite-care, etc., or a child who qualifies for free or reduced lunches from school). "High" SES was defined as not receiving free services.
  Participants
    Low SES | 36 | 42 | 78
    High SES | 20 | 14 | 34
    Prefer not to answer | 2 | 2 | 4
Sexual Orientation [Count of Participants; unit: Participants]
  Straight | 43 | 46 | 89
  LGBQ | 11 | 10 | 21
  Prefer not to answer | 4 | 2 | 6
The Revised Conflict Tactics Scales (CTS-2) [Mean (Standard Deviation); unit: units on a scale] — The Physical Assault subscale of the Conflict Tactics Scale (CTS-2), developed by Straus et al. (1996), was used to analyze changes in past-two-month peer violence in iDOVE participants, relative to an automated health-and-safety brief intervention and text message program. There are 14 items that measure violent behavior, each scored based on how frequently the participant has experienced the behavior (0=never to 6=20+ times). Score is summed, so the minimum score possible is 14*0=0 (lowest level of violence) and the maximum score possible is 14*6=84 (highest level of violence).
  units on a scale | 5.07 (6.72) | 2.69 (2.64) | 3.88 (5.22)
The Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) is a 9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression based on diagnostic criteria of depression from the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV. It asks about the patient's experience in the last 2 weeks. Responses range from "0" (Not at all) to "3" (nearly every day). The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. A total of 10 or above is suggestive of the presence of depression.
  units on a scale | 9.43 (3.82) | 8.78 (3.49) | 9.10 (3.66)
The Beck Depression Inventory (BDI-2) [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI-2) is a 1996 revision of the BDI, developed in response to the DSM-IV, which changed many of the diagnostic criteria for Major Depressive Disorder. Participants were asked to rate how they have been feeling for the past two weeks. It contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
  units on a scale | 13.60 (8.59) | 13.41 (10.10) | 13.51 (9.33)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms
Description: Becks Depression Inventory (BDI-2): To analyze changes in past-two-week depressive symptoms in iDOVE participants, relative to an automated health-and-safety brief intervention and text message program. The Beck Depression Inventory (BDI-2) is a 1996 revision of the BDI, developed in response to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV, which changed many of the diagnostic criteria for Major Depressive Disorder. Participants were asked to rate how they have been feeling for the past two weeks. It contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Time Frame: Enrollment, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment (8 wks after close of intervention)
Population: Stratified by baseline "moderate depressive symptoms" (BDI>=20).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- iDOVE Intervention (ED+Text): 1. In-ED brief session, introducing basic principles of cognitive behavioral theory (CBT) and the structure of the text-message portion of the intervention
  2. Eight-week longitudinal tailored CBT-based text-message program
  iDOVE Intervention (ED+text): 1) In-ED brief session, introducing basic principles of cognitive behavioral theory (CBT) and the structure of the text-message portion of the intervention 2) Eight-week longitudinal tailored text-message program
- Control (EUC): 1. In-ED brief session, discussing home safety & nutrition
  2. Eight-week longitudinal home safety & nutrition text-message program
  Control (Enhanced Usual Care (EUC)): 1) In-ED brief session, discussing home safety & nutrition 2) Eight-week longitudinal home safety & nutrition text-message program
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
Number analyzed (Participants) | 58 | 58
units on a scale
  BDI Score: Baseline | 13.6 (8.6) | 13.4 (10.1)
  BDI Score: 8 week | 14.8 (12.4) | 15.0 (11.9)
  BDI Score: 16 week | 12.5 (12.8) | 11.7 (11.0)
  BDI Score where baseline >=20: Baseline: number analyzed (Participants) | 16 | 15
  BDI Score where baseline >=20: Baseline | 24.5 (4.2) | 27.9 (9.2)
  BDI Score where baseline >=20: 8 week: number analyzed (Participants) | 16 | 15
  BDI Score where baseline >=20: 8 week | 19.9 (12.1) | 27.2 (11.5)
  BDI Score where baseline >=20: 16 week: number analyzed (Participants) | 16 | 15
  BDI Score where baseline >=20: 16 week | 21.9 (14.9) | 25.2 (10.0)
Statistical Analysis 1: Comparison: iDOVE Intervention (ED+Text) vs Control (EUC); BDI Score where baseline >=20: 8 week; Test type: Superiority; p = 0.07, Mixed effects longitudinal regression; Mean Difference (Final Values) = -7.48, Standard Error of Mean 4.11 — d=0.37

2. Primary Outcome: Change in Peer Violence Involvement
Description: The Physical Assault subscale of the Conflict Tactics Scale (CTS-2), developed by Straus et al. (1996), was used to analyze changes in past-two-month peer violence in iDOVE participants, relative to an automated health-and-safety brief intervention and text message program. There are 14 items that measure violent behavior, each scored based on how frequently the participant has experienced the behavior (0=never to 6=20+ times). Score is summed, so the minimum score possible is 14*0=0 (lowest level of violence) and the maximum score possible is 14*6=84 (highest level of violence).
Time Frame: as for outcome 1
Population: Stratified by higher baseline violence (CTS score >=4)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
Number analyzed (Participants) | 58 | 58
units on a scale
  CTS Score: Baseline | 3.0 [0.0 to 36.0] | 2.0 [0.0 to 9.0]
  CTS Score: 8 week | 2.5 [0.0 to 29.0] | 3.0 [0.0 to 15.0]
  CTS Score: 16 week | 2.0 [0.0 to 29.0] | 1.0 [0.0 to 32.0]
  CTS Score where baseline >=4: Baseline: number analyzed (Participants) | 24 | 18
  CTS Score where baseline >=4: Baseline | 8.0 [0.0 to 32.0] | 6.5 [0.0 to 15.0]
  CTS Score where baseline >=4: 8 week: number analyzed (Participants) | 24 | 18
  CTS Score where baseline >=4: 8 week | 4.0 [0.0 to 27.0] | 4.0 [0.0 to 14.0]
  CTS Score where baseline >=4: 16 week: number analyzed (Participants) | 24 | 18
  CTS Score where baseline >=4: 16 week | 2.0 [0.0 to 29.0] | 5.0 [0.0 to 32.0]
Statistical Analysis 1: Comparison: iDOVE Intervention (ED+Text) vs Control (EUC); CTS Score where baseline >=4: 8 week; Test type: Superiority; p = 0.01, quantile regression models; Controlled for baseline and gender; Median Difference (Final Values) = -7.29, Standard Error of Mean 2.62 — d=0.46

3. Secondary Outcome: Acceptability/Feasibility: Follow Up Rate
Description: Retention Rate: % of consented participants who completed follow up
Time Frame: 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment (8 wks after close of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
Number analyzed (Participants) | 58 | 58
Participants
  8 week follow up | 55 | 55
  16 week follow up | 54 | 52

4. Secondary Outcome: Acceptability/Feasibility: Engagement of Intervention Group
Description: Among the intervention group, how many participants responded to at least one of the daily text message queries, and how many requested on-demand support text-messages.
Time Frame: Enrollment to 16 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | iDOVE Intervention (ED+Text)
Number analyzed (Participants) | 58
Participants
  Responded to >=1 of the daily mood queries | 56
  Requested on-demand support text-messages | 22

5. Secondary Outcome: Acceptability/Feasibility: Participant Satisfaction
Description: The Customer Satisfaction Questionnaire (CSQ-8) developed by Larsen et al. (1979) is an 8-item survey where each item is scored 1 (poor) to 4 (excellent). It is scored by summing the individual item scores to produce a range of 8 to 32, with high scores indicating greater satisfaction.
Time Frame: 8 weeks post-enrollment (close of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
Number analyzed (Participants) | 58 | 58
units on a scale | 32.3 (5.7) | 31.2 (5.5)
Statistical Analysis 1: Comparison: iDOVE Intervention (ED+Text) vs Control (EUC); Test type: Superiority; p = 0.33, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through study completion (2 years)
Arm/Group | iDOVE Intervention (ED+Text) | Control (EUC)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

LIMITATIONS AND CAVEATS:
1. This study was not adequately powered to show efficacy.
2. This study enrolled during a convenience sample of shifts, at a single ED, excluding non-English-speaking adolescents; these limitations may introduce bias or reduce generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02332239/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT02332239/Prot_SAP_001.pdf